CLINICAL TRIAL: NCT03177304
Title: Web Based Therapist Training in Interpersonal Psychotherapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Psychological Consultation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R43MH106169 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Depression
Keywords: Interpersonal Psychotherapy; Internet; Training; Depression; Dissemination
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web based IPT Training (Experimental): All subjects (trainees) received the web based training, consisting of an on-line tutorial, remote live training via videoconferencing, and access to a post-training web portal
  Interventions: Other: Web based IPT Training

INTERVENTIONS:
Other: Web based IPT Training

SUMMARY:
The National Institutes of Mental Health has identified the use of empirically based mental health treatments (i.e., treatments with research supporting efficacy) as a priority, yet there is a shortage of clinicians trained in these approaches. This study develops an on-line therapist training program for Interpersonal Psychotherapy (IPT), a particularly well-researched yet particularly little disseminated, empirically based treatment, in order to facilitate wider dissemination of this approach.

DETAILED DESCRIPTION:
Experts from scientific, ethical, and economic perspectives have stressed the need for evidence-based mental health treatments, i.e., 'treatment based on the best available science or research evidence.' While several evidence-based treatments have been developed, there is a critical shortage of clinicians trained in these approaches. NIMH has identified the dissemination and implementation of evidence-based interventions as a top priority. One of the best studied evidence-based psychological treatments is interpersonal psychotherapy (IPT). Several decades of clinical trials have documented the efficacy of IPT across a diversity of mental health disorders and demonstrated the feasibility of teaching IPT to therapists from a range of backgrounds. Unfortunately, relatively few clinicians have been trained in IPT; as a result, few patients benefit from this treatment. The long term objective of this project is to meaningfully increase the number of mental health professionals trained in IPT by developing a set of internet training tools which will facilitate widespread dissemination of this training. In contrast to other evidence based therapies (e.g., cognitive behavior therapy), for which new training technologies have now been extensively studied, limited efforts to disseminate IPT to date have relied on traditional approaches (e.g., workshops), which are not cost-effective or easily accessible. In phase we will develop a prototype IPT training program and test its feasibility and efficacy. The training will comprise three components: a) An on-line, interactive, multi-media tutorial presenting the principles, stages, and techniques of IPT, b) Live, applied clinical training using videoconferencing in order to hone and evaluate trainees' clinical skills in IPT, and c) An on-line portal (IPT Case Tracker) to help therapists maintain adherence and facilitate integration of IPT into their ongoing clinical practice. Twenty-four clinicians from various mental health disciplines without prior IPT training will be recruited. Trainees will be tested on their knowledge of IPT concepts before and after completing the tutorial. Following completion of the tutorial, trainees will conduct an IPT session with a standardized patient while being observed by the trainer in real time using videoconferencing, in order to transfer knowledge into applied skills. After completing training, trainees will utilize the internet portal to help incorporate IPT into their clinical practice. The interactive portal will prompt trainees with brief reminders before IPT sessions and will administer a post-session checklist to help maintain and to monitor ongoing adherence to IPT. Feasibility and user satisfaction for the tutorial, live training and internet portal will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Practicing clinicians treating adult depressed patients

Exclusion Criteria:

* Able to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change on Test on IPT Concepts | change baseline and one month
  38-item test on knowledge of IPT concepts and skills

IPD SHARING:
Plan to Share IPD: No